CLINICAL TRIAL: NCT03123016
Title: A Split Body Study of the Effects of Combined Therapy With Narrow-Band Ultraviolet B Phototherapy and Apremilast for the Treatment of Vitiligo
Brief Title: Combined Therapy With Narrow-Band Ultraviolet B Phototherapy and Apremilast for the Treatment of Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Mark Lebwohl, Professor and System Chair, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-1261
Record Dates: First submitted 2017-04-11; First posted 2017-04-21 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Vitiligo
Keywords: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomized to treatment with narrowband UVB two to three times weekly to one half of their body for a total of 16 weeks, while the contralateral side of the body is covered by a special garment to prevent any UVB treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vitiligo with Apremilast and NB-UVB phototherapy (Experimental): Each participant will be compared with one side of the body to the other side
  Interventions: Drug: Apremilast; Procedure: NB-UVB phototherapy

INTERVENTIONS:
Drug: Apremilast — Apremilast 30 mg orally, twice daily. (oral tablet)
Procedure: NB-UVB phototherapy — treatment with narrowband UVB two to three times weekly to one half of their body for a total of 16 weeks

SUMMARY:
Vitiligo is a common acquired disorder of pigmentation affecting 0.5% to 1% of the world population. Sharply demarcated patches of depigmentation, which can affect all ethnicities, and can lead to cosmetic disfiguration and psychosocial distress, characterize the disease. The etiology of vitiligo remains unknown. Various mechanisms have been proposed, such as autoimmunity, self-destruction, biochemical, genetic, neural, oxidative stress, and an imbalance of epidermal cytokines leading to inflammation and selective loss of epidermal melanocytes. Currently, the most popular theory is autoimmunity. Previous studies noted that around 25-30% of patients have at least one other autoimmune disease, such as autoimmune thyroid disease, Addison's disease, pernicious anemia, and alopecia areata. Currently, NB-UVB phototherapy is the most widely used therapeutic option for vitiligo affecting more than 10-20% of the skin surface, as it is generally considered to be a safe initial treatment. Potential side effects include phototoxic reaction, thickening of the skin and koebnerization. NB-UVB is a band of UV radiation with a wavelength of 311-313 nm. UVB induces mitogenesis and migration in melanocytes mediated by several factors such as IL-1, TNF alpha, and leukotriene C4. UV radiation produces increased number and activity of melanocytes, increased melanin density, elongation and branching of dendrites, with increased transfer of more heavily melanized melanosomes to keratinocytes, seen clinically as increased pigmentation. Apremilast is an oral small molecule phosphodiesterase-4 (PDE4) inhibitor that has been shown to regulate inflammatory mediators. Apremilast enters cells by passive diffusion and, once intracellular, binds PDE4. PDE-4, the dominant phosphodiesterase expressed in immune cells, degrades cyclic AMP (cAMP) into AMP. PDE4 inhibition thereby elevates intracellular cAMP, which can down-regulate the inflammatory responses such as TNF-α, IFN-γ, interleukins (IL) 2, 12 and 23 through mechanisms such as partially inhibiting expression of inflammatory cytokines and increasing expression of anti-inflammatory mediators such as IL2 and IL10. The hypothesis is that apremilast will shut down the inflammatory insult in vitiligo and NB-UVB phototherapy will then be able to regenerate melanocytes and their activity. By examination of skin biopsies taken pre- and post-therapy, the study team aims to assess changes in immune and cellular markers in affected skin.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ≥ 18 years of age at the time of signing the informed consent document.
* Must be in general good health (except vitiligo) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
* Able to adhere to the study visit schedule and other protocol requirements.
* Subjects must be clinically diagnosed by the investigator to have at least 20% body surface area involvement of generalized type vitiligo.
* Fitzpatrick skin phototypes IV, V, and VI.
* Must meet the following laboratory criteria

  1. White blood cell count ≥ 3000/mm3 (≥ 3.0 x 109/L) and < 14,000/mm3 (< 14 x 109/L).
  2. Platelet count ≥ 100,000/μL (≥ 100 x 109/L).
  3. Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L).
  4. AST (SGOT) and ALT (SGPT) ≤ 2 x upper limit of normal (ULN). If the initial test shows ALT or AST > 2 times the ULN, one repeat test is allowed during the Screening Phase.
  5. Total bilirubin ≤ 2 mg/dL (34 μmol/L). If the initial test shows total bilirubin > 2 mg/dL (34 μmol/L), one repeat test is allowed during the Screening Phase.
  6. Hemoglobin ≥ 10 g/dL (≥ 6.2 mmol/L).
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; or

Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).

* Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product.

Exclusion Criteria:

* Clinically significant (as determined by the investigator) cardiac, endocrine, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, or immunologic disease, or other major uncontrolled diseases that will affect the health of the subject during the study or interfere with the interpretation of study results.
* Hepatitis B surface antigen positive at Screening (Visit 1).
* Hepatitis C antibody positive at Screening (Visit 1).
* History of positive human immunodeficiency virus (HIV), or congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency [CVID]). Active TB or a history of inadequately treated TB.
* Active substance abuse or a history of substance abuse within six months prior to Screening.
* Pregnant or breast feeding.
* History of allergy to any component of the IP.
* Major surgery within eight weeks prior to Screening (Visit 1) and/or planned surgery during the length of the study.
* Malignancy or history of malignancy, except for:

  1. treated (ie, cured) basal cell or squamous cell in situ skin carcinomas;
  2. treated (ie, cured) cervical intraepithelial neoplasia (CIN) or carcinoma in situ of the cervix with no evidence of recurrence within 5 years prior to Screening (Visit 1).
* Unstable asthma (eg, acute episodes of exacerbation [nocturnal episodes, sudden episodes triggered by unidentifiable factors] despite a stable regimen of anti-asthmatic medications); prior episode(s) of life-threatening asthma; or asthma that requires inhaled budesonide or equivalent at >1200 μg/day or fluticasone propionate at > 880 μg/day along with another anti-asthmatic drug such as a long-acting beta-agonist.
* A history of and/or concurrent condition of serious hypersensitivity (eg, anaphylaxis) to drugs, foods, or other allergens without access to emergency rescue medication such as epinephrine.
* Persistent or recurring bacterial infection requiring systemic antibiotics, or clinically significant viral or fungal infections, within two weeks of Screening (Visit 1). Any treatment for such infections must have been completed at least two weeks prior to the Screening Visit and no new/recurrent infections should have occurred prior to the Baseline Visit.
* Active skin infection requiring systemic antimicrobials at Baseline/Randomization (Visit 2).
* Skin lesion(s) due to conditions other than vitiligo that would interfere with the study specified assessments.
* Prior treatment with apremilast, or participation in a clinical study involving apremilast.
* Use of phototherapy (ie, UVB, UVA) or systemic immunosuppressive drugs (including, but not limited to, cyclosporine, corticosteroids, mycophenolate mofetil, azathioprine, Methotrexate, or tacrolimus), or oral preparations of herbal immunomodulatory medications within four weeks prior to Baseline/Randomization (Visit 2).
* Use of interferon-γ within 12 weeks prior to Baseline/Randomization (Visit 2).
* Use of abatacept, adalimumab, certolizumab pegol, etanercept, golimumab, infliximab, or tocilizumab within 12 weeks prior to Baseline/Randomization (Visit 2).
* Use of oral janus kinase (JAK) inhibitors (e.g. tofacitinib, ruxolitinib) within 12 weeks prior to Baseline/Randomization (Visit 2).
* Use of omalizumab, rituximab, ustekinumab, alefacept, briakinumab, or other therapeutic antibody products within 24 weeks prior to Baseline/Randomization (Visit 2).
* Use of any investigational drug within four weeks or five PK or PD half lives (whichever is longer) prior to Baseline/Randomization (Visit 2).
* Use of topical corticosteroid preparations, topical calcineurin inhibitors, or other topical preparations with immunomodulatory properties within 2 weeks prior to Baseline/Randomization (Visit 2).
* Prior history of suicide attempt at any time in the subject's lifetime prior to Baseline (Visit 2) or major psychiatric illness requiring hospitalization within 3 years prior to Baseline (Visit 2).
* Prolonged sun exposure or use of tanning booths, which may confound the ability to interpret data from the study.
* Subjects whose vitiligo has not responded to at least 6 months of treatment with NB-UVB.
* Subjects with segmental or localized vitiligo.
* Subjects with a history of therapeutic attempts at depigmentation.
* Fitzpatrick skin phototypes I, II, and III
* Subjects with history of photosensitivity ⁄ photo exaggerated dermatoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Change in proportion of responders to treatment from Week 16 to Week 32 | Week 16 and Week 32
  The proportion of responders to apremilast plus concomitant NB-UVB at week 32 compared to the proportion of responders to NB-UVB phototherapy at week 16.

SECONDARY OUTCOMES:
Body Surface Area (BSA) | Week 32 and Week 48
  One hand unit, which encompasses the palm plus the volar surface of all the digits, is approximately 1% of the total body surface area and is used as a guide to estimate each body region.
VASI score - Vitiligo Area and Severity Index (VASI) | Week 32 and Week 48
  One hand unit, which encompasses the palm plus the volar surface of all the digits, is approximately 1% of the total body surface area and is used as a guide to estimate the baseline percentage of vitiligo involvement in each body region. The body is divided into five separate and mutually exclusive regions: hands, upper extremities (excluding hands), trunk, lower extremities (excluding feet), and feet. The axillary region is included with the upper extremities while the buttocks and inguinal areas are included with the lower extremities. The extent of residual depigmentation is expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%. At 100% depigmentation, no pigment is present; at 90%, specks of pigment are present; at 75%, the depigmented area exceeds the pigmented area; at 50%, the depigmented and pigmented areas are equal; at 25%, the pigmented area exceeds the depigmented area; at 10%, only specks of depigmentation are present.
VETF score - Vitiligo European Task Force (VETF) score | Up to 64 weeks
  The VETF is a validated scoring system that assesses 3 dimensions of the disease (extent, staging, and spreading/progression). (1) the extent of vitiligo will be estimated as the percentage of vitiligo involvement of 5 body sites. (2) Stage of vitiligo will be assessed as 0 (normal pigmentation), 1 (incomplete depigmentation), 2 (complete depigmentation), 3 (partial hair whitening [<30%]), and 4 (complete hair whitening). (3) Spreading of vitiligo will be scored as 0 (stable disease), -1 (observed ongoing subclinical repigmentation), and +1 (additional patches in a given area or observed ongoing subclinical depigmentation). The VETF score calculated as follows:
  VETF Extent or Staging or Spreading = Sum of all specific values for that category from all body sites (% of Area affected for Extent; 0-20 for Staging; -5 to +5 for Spreading).
Dermatology Life Quality Index | Up to 64 weeks
  The DLQI is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions, and its use has been described in over 1000 publications including many multinational studies. The DLQI is the most frequently used instrument in studies of randomized controlled trials in dermatology.
Visual Analogue Scale (VAS) | Up to 64 weeks
  The VAS is commonly used as the outcome measure in research studies. A VAS for satisfaction is a horizontal line of 100-mm long. At the beginning and at the end, there are two descriptors representing extremes of satisfaction (i.e. no satisfaction and extreme satisfaction). The patients rate their satisfaction by making a vertical mark on the 100-mm line. The measurement in millimeters is converted to the same number of points ranging from 0 to 100 points. The exact question will be "Are you satisfied with your study treatment?"
Number of Adverse Events | Up to 64 weeks
  Safety analyses will be performed on the safety population. Safety will be evaluated by tabulations of adverse events (AEs) and will be presented with descriptive statistics at each visit. AEs will be coded using the CTCAE, Common Terminology Criteria for Adverse Events, V 4.0. The CTCAE v4.0 AE terms are MedDRA's LLTs (Lowest Level Terms) which are based on their MedDRA (System Organ Class). The number and percentage of subjects experiencing an AE/SAE will be stratified by system organ class, or a preferred term, and/or severity of the adverse event, and recorded and tabulated overall.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No